CLINICAL TRIAL: NCT02163655
Title: Effectiveness of Postpartum Furosemide on Recovery Blood Pressure in Puerperal Women with Severe Preeclampsia: a Randomized Clinical Trial
Brief Title: Diuretics for Postpartum High Blood Pressure in Preeclampsia
Acronym: DIUPRE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Principal Investigator, Leila Katz, PhD, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DIUPRE; DIUPRE (Other: Brazil Ministry of Health)
Record Dates: First submitted 2014-06-09; First posted 2014-06-13 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2021-07

CONDITIONS: Preeclampsia
Keywords: preeclampsia, very high blood pressure, diuretics
MeSH Terms: conditions — Pre-Eclampsia | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PLACEBO (Placebo Comparator): PLACEBO: placebo, oral, every 24 hours for maximum 5 days
  Interventions: Drug: Placebo
- FUROSEMIDE (Experimental): FUROSEMIDE: 20mg furosemide, oral, every 24 hours for maximum 5 days
  Interventions: Drug: FUROSEMIDE

INTERVENTIONS:
Drug: FUROSEMIDE — Furosemide, 20mg pills, will be administered every 24 houras, for a maximum of five days
  Other Names: Lasix
  Arms: FUROSEMIDE
Drug: Placebo — Placebo pills, identical to the intervention (furosemide pills), will be administered every 24 hour for a maximum of five days
  Arms: PLACEBO

SUMMARY:
The purpose of this study is to determine if furosemide administered after the first 24 hours of delivery, in women with severe peeclampsia and eclampsia accelerates high blood pressure control and diminishes hospital stay.

DETAILED DESCRIPTION:
A placebo-controlled study that will be conducted including 120 postpartum women with severe preeclampsia . Women who are previosuly diuretic users, with renal impairment, hemodynamic instability or with contraindications to diuretic use will be excluded. Informed consent will be obtained from all participants . Patients will be randomized to receive furosemide ( 40mg orally every twenty-four hours ) or placebo for maximum of five days. The variables are systolic and diastolic blood pressure, frequency of very high blood pressure, need for maintenance of antihypertensive therapy , number of antihypertensive agents used to control blood pressure , urine output , length of hospital stay , adverse effects and maternal complications . Except for the study drug, patients will receive all care and monitoring according to the hospital protocol and decision to initiate or modify antihypertensive therapy will be defined by the attending physician, as well as the decision to discharge. If the patient is discharged before five days of the protocol drug, this drug will be stopped. Teh patients may decide to leave the study at any moment. Data will be collected by researches daily. Plan statistical analysis will be performed using the public domain program Epi Info 7.0 and the mean and dispersion measures for numerical variables will be calculated. To compare means obtained every day and between groups will be used analysis of variance ( ANOVA ) . Nominal variables were compared using the X2 test or Fisher if necessary. Be considered significant at p < 0,05. The risk ratio (RR) is calculated as a measure of the relative risk for the different outcomes , according to furosemide or placebo

ELIGIBILITY:
Inclusion Criteria:

* Preeclampsia
* Urine output > 50ml/h
* End of postpartum magnesium sulphate

Exclusion Criteria:

* Cronic hypertension
* Bloor pressure < 140mmHg and < 90mmHg
* Diuretic use
* Renal impairment
* Diabetes, sickle cell disease ou rheumatologic disease
* Hemodinamic instability
* Potassium < 3mEq/L
* Contraindications for fusoremide use

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-06-20 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Mean blood pressure | from 24 hours after delivery to first 15 days of delivery

SECONDARY OUTCOMES:
postpartum hospital stay | from 24 hours after delivery to 15 days
  Time until discharge of the hospital
Maintenance of antihypertensive therapy | From 24 hours up to 15 days of delivery
  Number of antihypertensive agents used to control blood pressure at hospital discharge; time elapsed to control blood pressure; daily urine output; reduction of edema; length of hospital stay; frequency of adverse effects: hypokalemia, polydipsia, headache, mental confusion, muscle pain, tetany, muscle weakness, heart rhythm disturbances and gastrointestinal symptoms; frequency of maternal complications: imminent eclampsia, eclampsia, infection, bleeding manifestations, shock and maternal death.
frequency of adverse effects | From 24 hours to 15 days after delivery
  Presence of hypokalemia, polydipsia, headache, mental confusion, muscle pain, tetany, muscle weakness, heart rhythm disturbances and gastrointestinal symptoms;
frequency of maternal complications | From 24 hours up to 15 days after delivery
  Frequency of imminent eclampsia, eclampsia, infection, bleeding manifestations, shock and maternal death.

OTHER OUTCOMES:
Frequency of very high blood pressure episode | from 24 hours after delivery until 15 days after delivery
  Frequency of very high blood pressure (Systolic blood pressure >180mmHg and diastolic blood pressure >110mmHg) episodes
Blood pressure control | From 24 hours after delivery to 15 days
  Absence pf very blood pressure episodes in 24 hours period

CONTACTS AND LOCATIONS:
Overall Officials: Leila Katz, MD PhD, Study Director — IMIP
Locations (1):
- IMIP, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Cursino T, Katz L, Coutinho I, Amorim M. Diuretics vs. placebo for postpartum blood pressure control in preeclampsia (DIUPRE): a randomized clinical trial. Reprod Health. 2015 Aug 5;12:66. doi: 10.1186/s12978-015-0057-0. PMID 26242730